CLINICAL TRIAL: NCT06962722
Title: The Effect of Upper Limb Low-intensity Motor Control Training (uMCON) Program on Cognitive Function in Healthy Older Adults: A Pilot Study
Brief Title: The Effect of Upper Limb Low-intensity Motor Control Training Program on Cognitive Function in Healthy Older Adults
Acronym: uMCON
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Bethan Phillips, Professor, University of Nottingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: FMHS 331-0723
Record Dates: First submitted 2024-09-27; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Cognitive Impairment
Keywords: neuromuscular training; older adults; cognitive impairment; exercise
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention Group (Experimental): uMCON training group
  Interventions: Other: Upper limb motor control training (uMCON)

INTERVENTIONS:
Other: Upper limb motor control training (uMCON) — The exercise program protocol was determined using elbow flexion (Biceps brachii) and elbow extension (Triceps) on a special platform developed for the arm. In this computer-based exercise, participants are asked to follow a small ball on the screen in different lines at certain percentages of maximum muscle strength (10%, 25%, 50%, and so on). Neuromuscular training will be worked on with this exercise.

SUMMARY:
This healthy volunteer intervention study is designed to evaluate the effectiveness of upper limb motor control training (uMCT) on physical and cognitive functions in older adults. The primary objectives of the study are twofold:

Assess the Impact on Physical and Neuromuscular Function: The study seeks to determine whether uMCT positively influences physical performance, including motor coordination and neuromuscular function, in older adults.

Assessment the Impact on Cognitive Function: The study aims to investigate whether uMCT enhances cognitive abilities in older adults.

In addition to these main goals, the study will also assess the feasibility and safety of implementing uMCT in an older adult population.

The main questions it aims to answer are:

Does uMCON training have a positive effect on physical function and neuromuscular function in older adults?

Does uMCON training have a positive effect on cognitive function in older adults? The researchers designed this study to show whether uMCON training works on physical function (balance, gait, and so on) and cognition in older adults.

Participants will come to Derby Royal Hospital Medical School to attend uMCON training three days a week for 1 month. They will attend pre-training, post-training, and follow-up (after 1 month) control assessment sessions.

DETAILED DESCRIPTION:
Experimental protocol

Participants:

This study will be carried out on 24 healthy participants (aged between 65-85 years), with an aim to recruit 50% males. Participants will be randomised (via sealed envelope) to the uMCT group or a no-intervention control group (PPI). Before enrolment on to the study, participants will complete a screening session which will include an electrocardiogram (ECG), blood pressure check, and general health questions, including previous medical history. This session will also provide potential participants an opportunity to ask any questions about the study that they may have after reading the participant information sheet (PIS). If an abnormal screening result is encountered, this will be discussed with the participant and their GP will be informed in writing. All participants will be informed in detail about the procedures and risks of the study via the PIS and the opportunity to ask questions, before their written informed consent is obtained.

Assessment sessions:

All participants will be requested to attend 3 assessment sessions, in addition to 4-weeks uMCT (3x/wk) for the intervention group. For participants in the PPI group (no intervention control group), they will also attend the research unit 3x/wk to participate in patient and public involvement (PPI) (in research) activities. These actives will include, as examples, discussion around the importance/relevance of upcoming studies, lay review of participant/patient facing documents, assistance with research dissemination. Given the primary endpoint of this study is cognition, this approach will mitigate the impact of any adaptation in the uMCT group being due to their regular in-person engagement with the research team as all participants will have this. It will also allow participants in the no-intervention group to feel that their time is productive and worthwhile.

The assessment sessions will take place:

* before the intervention (V1),
* after the 4-week intervention (V2),
* and after 4-weeks de-training (V3) to determine any adaptation retention.

Each of these sessions will be identical and will comprise:PPI

* Evaluation of cognitive function using MOCA, TMT and SCWT,
* The nine-hole Peg Test to determine dexterity,
* Isometric dynamometery to determine MVC for elbow flexion and knee extension (to assess non-joint specific adaptation),
* Surface electromyography (sEMG) of the triceps brachii and intramusculer electromyography (iEMG) of vastus lateralis to determine muscle activation patterns (training specific and non-specific),
* Simple (eyes open) and complex (eyes closed) balance tests,
* Timed Up-and-Go (TUG) to determine mobility,
* The Short Physcial Performace Battery (SPPB) to assess overall physical performance.

Each assessment session is expected to last a maximum of 3 hours, allowing sufficient time for explanation of each component at each visit.

Training Sessions:

uMCT will involve 3 sessions each week for 4 weeks based on elbow flexion. Each session will last ~20 minutes and will be fully supervised by a member of the research team. During each training session, participants will be asked to follow a sinusoidal force line on a screen by contracting their elbow flexors. Six to 10 different force tracking wave forms will be performed in each session at 10%, 25%, or 40% of MVC with an amplitude of ±2%, ±4%, or ±8%. Each wave form will last 20-30 seconds with 60 seconds of rest between each.

ELIGIBILITY:
Inclusion Criteria:

* • Willing and able to give informed consent for participation in the study

  * Aged between 65-85 years

Exclusion Criteria:

* • Diagnosis of cognitive impairment

  * Current or recent (<5y) malignancy
  * History of or current psychiatric illness
  * History of or current neurological condition (e.g., epilepsy, Parkinsons disease, cerebrovascular disease)
  * Severe respiratory disease (e.g., uncontrolled asthma, COPD, pulmonary hypertension)
  * Active cardiovascular disease: Uncontrolled hypertension (BP>160/100mmHg); Recent (<12mo) cardiac event; Heart failure (Class III/IV); Significant arrhythmia; Unstable angina
  * Metabolic disease: Untreated hyper/hypo-parathyroidism; Cushing's disease; Type 1 or 2 diabetes
  * Significant musculoskeletal disorders (based on clinical opinion)
  * Family history of early (<55y) death from cardiovascular disease

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Outcome Measure Title: Rate of participants whose cognition improved with upper limb motor control training. | Baseline, 4 week, and 8 week
  Number of Participants: 20 Control group: No Rate of Female/Male: 50%/ 50% Time frame: 1 month upper limb neuromuscular training Assessment time: Pre-training, Post-training, Follow-up(after 4 weeks) Cognition questionnaire is used (MOCA).

SECONDARY OUTCOMES:
Clinically relevant functional outcomes (motor control, strength, dexterity, overall physical function) | Baseline, 4 week, and 8 week
  * The nine-hole Peg Test to determine dexterity,
  * Isometric dynamometery to determine MVC for elbow flexion and knee extension (to assess non-joint specific adaptation),
  * Surface electromyography (sEMG) of the triceps brachii and intramusculer electromyography (iEMG) of vastus lateralis to determine muscle activation patterns (training specific and non-specific),
  * Simple (eyes open) and complex (eyes closed) balance tests,
  * Timed Up-and-Go (TUG) to determine mobility,
  * The Short Physcial Performace Battery (SPPB) to assess overall physical performance.
Plasma pro/anti-inflammatory cytokine levels | Baseline, 4 week, and 8 week
  Only a single blood sample (<10ml) will be taken from participants at each assessment session via venepuncture. This will only be performed by an individual trained and competent in this technique. Blood samples will be centrifuged, and plasma stored at -20 to -80 degrees until batch-analysis at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Sirin Ekici, PhD, Study Director — The University of Nottingham; Mehmet C Yildirim, PhD, Study Director — The University of Nottingham
Locations (1):
- The University of Nottingham Medical School, Derby, Derbyshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Access to personal (identifiable) information is limited only to research staff involved in the participation elements of this study, and to audit staff as detailed above.